CLINICAL TRIAL: NCT04416516
Title: A Phase 2A Study to Assess the Safety and Efficacy of ASN-002 Combined With a Hedgehog Pathway Inhibitor in the Treatment of Multiple Low Risk Basal Cell Carcinomas in Sporadic or Basal Cell Nevus Syndrome Patients
Brief Title: Safety and Efficacy of ASN-002 Combined With a Hedgehog Pathway Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascend Biopharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASN-002-003
Record Dates: First submitted 2020-05-21; First posted 2020-06-04 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Basal Cell Carcinoma; Basal Cell Nevus Syndrome
Keywords: high frequency basal cell carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome | interventions — gusacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1, Patients with 1 Tumour (Experimental): Participants with 1 Target Tumour will receive 3 x ASN-002 1.0x10(11) Injections
  + VISMODEGIB (150 mg) daily for 4 weeks.
  Interventions: Biological: ASN-002
- Arm 2, Patients with 3 or more Tumours (Experimental): Participants with 3 or more Target Tumours will receive 3 x ASN-002 1.0x10(11) Injections (per tumour) + VISMODEGIB (150 mg) daily for 4 weeks.
  Interventions: Biological: ASN-002
- Arm 6 Patients with 3 or more Tumours (Experimental): Participants with 3 or more Target Tumours will receive 3 x ASN-002 1.5x10(11) Injections (per tumour) + VISMODEGIB (150 mg) daily for 4 weeks
  Interventions: Biological: ASN-002

INTERVENTIONS:
Biological: ASN-002 — ASN-002 has been designed for clinical applications, especially for intratumoral administration in the treatment of various cancers. This rAd vector delivers the gene of interest, in the case of ASN-002 the human IFNγ gene, into target cells. The rAd vector in ASN-002 is replication deficient and although it infects cells, it is not able to replicate in the tumor or in normal human cells. The infected cells are able to transcribe and translate the IFNγ DNA leading to a sustained local concentration of IFNγ in the tumor mass that is designed to avoid high levels of systemic IFNγ that may be lead to unacceptable toxicity.

SUMMARY:
The primary objectives are to:

1. Evaluate the safety and tolerability of intralesional ASN-002 when administered in combination with oral vismodegib in patients with Basal Cell Carcinomas (BCC)s;
2. Evaluate the efficacy of intralesional ASN-002 in target tumours when administered in combination with oral vismodegib in patients with BCCs.

The secondary objective is to:

1) Evaluate the efficacy of intralesional ASN-002 in non-target tumours when administered in combination with oral vismodegib in patients with BCCs.

The exploratory objective is to:

1) Evaluate immunological biomarkers during the course of treatment.

DETAILED DESCRIPTION:
Methodology:

This study will evaluate ASN-002 (in the dose range 0.5 to 1.5x10(11) vp/mL) with the Hh inhibitor vismodegib (Erivedge®). The study will initially evaluate two Arms receiving 1.0 x 10(11) vp/injection, and following a safety review, may implement further arms in an adaptive study design.

Following screening and baseline biopsies for target and non-target tumours, eligible subjects will be enrolled in the study.

Cycle 1: Treatment with vismodegib (daily dose of 150 mg) for 4 weeks and ASN-002 for 3 weeks (i.e., three ASN-002 injections in total):

* Day 1 to Day 14 - vismodegib alone
* Day 15 - vismodegib and ASN-002
* Day 16 to Day 21 - vismodegib alone
* Day 22 - vismodegib and ASN-002
* Day 23 to Day 28 - vismodegib alone
* Day 29 - ASN-002 alone

Clinical response will be assessed at Week 17, following which, the investigator may where clinically indicated, initiate Cycle 2.

Cycle 2: Treatment with vismodegib (daily dose of 150 mg) for 4 weeks, and one further injection with ASN-002:

* Day 1 to Day 7 - vismodegib alone
* Day 8 - vismodegib and ASN-002
* Day 9 to Day 28 - vismodegib alone

Surgical excision for all patients will occur between Week 25 and Week 33 at the investigators discretion, and dependent on when patient completed study treatment (1 or 2 treatment cycles). Up to 10 BCCs to be excised including 3 target tumours. Excisions can be conducted over 2 visits as per Investigator's discretion.

The Investigator may enrol eligible patients parallel into either Arm 1 or Arm 2, based on the number of tumours present. Up to 10 study BCC tumours (up to 3 target and up to 7 non-target) will be selected per patient.

Following review of at least Week 5 data for N=6 patients in Arm 1 and Arm 2, further Arms with varying doses of ASN-002 (in the dose range 0.5x10(11) vp or 1.5x10(11) vp) may be explored at the discretion of the Safety Review Committee (SRC). Vismodegib or ASN-002 may be evaluated as monotherapies to provide control groups to allow comparison of treatment Arms.

Safety and clinical assessments will be performed at Weeks 1, 3, 4, 5, 7, 17, 25 to 33.

Histological response will be evaluated in all study tumours via excision between Week 25 and Week 33 (as per investigator's discretion).

Six patients will be recruited to each Arm of the study, each Arm may be expanded to 12 patients at the discretion of the SRC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed previously untreated, BCC (nodular and superficial), 5-20 mm in maximum diameter, per the selection criteria for study BCC tumours. A punch biopsy (refer to study procedure manual for biopsy size selection) from the thickest part of all the target tumours is required for histological confirmation of BCC and to exclude BCC non-eligible subtypes.

   Note: If a patient has mix of nodular and superficial BCC tumours, at least one target tumour should be a nodular BCC.
2. Removal of < 25% of the area of each biopsied tumour by initial biopsy performed 1-12 weeks before Day 1. If the initial biopsy was performed >8 weeks prior to screening, the investigator may re-biopsy the tumour, provided not > 25% of the area of the original tumour is removed. Non-study tumours may be resected or treated at the discretion of the Investigator prior to study entry or if they develop during the study.
3. Hedgehog pathway inhibitor treatment naïve.
4. Acceptable general health as determined by the investigator, i.e. no serious or active medical or psychiatric illness or recreational or therapeutic drug or alcohol use that, in the opinion of the Investigator, would interfere with treatment, assessment or compliance with the protocol, ability to provide informed consent, or patient safety.
5. 18 years of age or older.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
7. Screening laboratory values as follows:

   1. Neutrophil count > 1500/mm3
   2. Haemoglobin > 9 g/dL
   3. Platelet count >100,000/mm3
   4. Prothrombin INR < 1.5
   5. Total bilirubin < 1.5 X upper limit of normal (ULN), except in the case of known Gilbert's syndrome
   6. Aspartate transaminase (AST), alanine transaminase (ALT) or alkaline phosphatase (ALP) < 2X ULN
   7. Creatinine < 1.5 X upper limit of normal (ULN)
8. Female patients who are documented infertile, postmenopausal for at least 1 year, surgically sterile or using acceptable and highly effective birth control for the duration of the study and for at least 3 months after last administration of the study treatments.
9. Male patients with female partners of child bearing potential, agreement to use two adequate contraception methods while being on vismodegib and for 3 months of completion. agreement not to donate semen for 3 months after completion of vismodegib.
10. Written informed consent prior to initiation of study-specified procedures.
11. Able and willing to comply with all study requirements, including surgical removal of tumour/tumour site at completion of study.
12. Baseline tissue sample adequate for determination of histological or other biomarkers.

Exclusion Criteria

1. Known or suspected metastatic disease or other active, invasive malignancy.
2. Female patients of childbearing potential who are lactating or pregnant (negative serum pregnancy test needed prior to dosing).
3. Clinically active or uncontrolled skin disease or tattoos that would interfere with evaluation of the area surrounding the target tumour (e.g. eczema, unstable psoriasis, xeroderma pigmentosa).
4. Known history of sensitivity to any of the ingredients in ASN-002 and any Hh pathway inhibitors.
5. Immunocompromised (e.g. known Hepatitis B or C infection, HIV infection) or receiving or expected to receive an immunomodulating agent (including immunosuppressive agents, cytotoxic drugs, biological agents, immunoglobulins, interferon or other immune or cytokine-based therapies. Use of inhaled or oral corticosteroids at doses higher than physiological replacement doses is an exclusion criterion).
6. Has received or is expected to receive treatment with psoralen plus UVA or UVB therapy within 6 months of the Screening visit.
7. Any prior systemic anti-tumour therapy or local treatment for target tumours prior to first dose.
8. History of immunological disorder, severe allergic reaction, moderate or severe asthma or known history of anaphylaxis or any other serious adverse reactions to any medication.
9. Any experimental or investigational agents within one month of first ASN-002 injection.
10. Any prior exposure to TG1041, TG1042 (ASN-002), any other adenoviral-based experimental agent, or any form of gene therapy within 6 months of first dose of vismodegib in the study.
11. Any prior exposure to vismodegib or any other Hh inhibitor within 6 months of first dose in the study.
12. Current therapy with any medications recognized to cause rhabdomyolysis or a prior history of rhabdomyolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Incidence of ASN-002 related Adverse Events in patients with previously untreated nBCC | Participants will be followed up to 6 months
  Incidence of Adverse Adverse events will be monitored
Microscopic clearance of the injected Target basal cell carcinoma. | Microscopic examinations of sample collected at weeks 25-33 after the first dose.
  Histological clearance (HC) will be defined as the absence of detectable evidence of BCC tumor cell nests in serial histological samples as determined by central pathology review.

SECONDARY OUTCOMES:
Microscopic clearance of the injected Non-Target basal cell carcinoma. | Microscopic examinations of sample collected at weeks 25-33 after the first dose.
  Histological clearance (HC) will be defined as the absence of detectable evidence of BCC tumor cell nests in serial histological samples as determined by central pathology review.

CONTACTS AND LOCATIONS:
Overall Officials: Clement Leong, Ph.D, Study Chair — Ascend Biopharmaceuticals Ltd; Gregory Siller, Principal Investigator — Central Brisbane Dermatology
Locations (7):
- Australia (7):
  - Central Brisbane Dermatology, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Veracity Clinical Research, Brisbane, Queensland
  - Sunshine Coast University Hospital, Sunshine Coast, Queensland
  - Sinclair Dermatology, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Burswood Dermatology, Perth, Western Australia